CLINICAL TRIAL: NCT02801006
Title: The Clinical Study of Silicone Hydrogel Daily Disposable Stenfilcon A Toric Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: JP-MKTG-201603
Record Dates: First submitted 2016-06-10; First posted 2016-06-15 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2017-12

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- stenfilcon A (Experimental): Participants will be randomized to wear stenfilcon A lens pair for two weeks during the cross over study.
  Interventions: Device: stenfilcon A
- etafilcon A (Active Comparator): Participants will be randomized to wear etafilcon A lens pair for two weeks during the cross over study.
  Interventions: Device: etafilcon A

INTERVENTIONS:
Device: stenfilcon A — contact lens
  Arms: stenfilcon A
Device: etafilcon A — contact lens
  Arms: etafilcon A

SUMMARY:
The aim of this study is to evaluate the clinical performance of stenfilcon A toric lenses compared with etafilcon A toric lenses for astigmatism. If it is valuable, the clinical performance of stenfilcon A toric lens is also evaluated compared with habitual lenses.

DETAILED DESCRIPTION:
This is a multi-sites, 50 subjects, randomized, open labeled, bilateral wear, dispensing study. Participants will be randomized to wear first lens pair for two weeks, and then crossover to second lens pair for two weeks.

ELIGIBILITY:
Inclusion Criteria:

A person is eligible for inclusion in the study if he/she:

* Is between 18 years of age and 42 years of age.
* Soft contact lens wearers who are not required to have Presbyopic correction.
* Soft contact lens wearers without trouble.
* Soft contact lens wearers who have the correctable astigmatism by lenses used in this study in the both eyes.
* Has a prescribed SCL (Soft Contact Lens) power within the range of powers of the SCL for astigmatism which is used in this study.
* Can achieve a corrected visual acuity of 1.0 or better.
* Can read and understand the study information document, and sign the participation consent form.
* Can visit the clinic at designated examination visits.
* Has received periodical examinations at an eye clinic within the past two years.

Exclusion Criteria:

A person will be excluded from the study if he/she:

* Has a systemic disease that may affect the ocular health.
* Is pregnant or lactating.
* Has received a systemic or local medication that may affect this study.
* Has an infectious eye disease.
* Has eye and systemic active allergic diseases that interferes with SCL wear.
* Has an eye disease which is clinically judged to be severe such as corneal vascularization, limbal hyperemia, and corneal epithelium disorder
* Has a history of hard contact lens wear within 30 days.
* Is currently participating in another clinical research study.
* Has undergone refractive surgery.

Ages: 18 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2016-04; Primary Completion 2016-06 (Actual); Study Completion 2016-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuji Kodama, MD, PhD, Principal Investigator — Director, Kodama Eye Clinic
Locations (2):
- Japan (2):
  - Kodama Eye Clinic, Terada, Kyoto
  - Dougenzaka Ioti Eye Clinic, Shibuya City, Tokyo-to

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: EYES
Groups:
- Stenfilcon A First, Then Etafilcon A; Etafilcon A First, Then Stenfilcon A: Participants randomized to wear stenfilcon A toric lens pair for two weeks then etafilcon A toric lens pair in the cross over study.
Period: Lens 1
Arm/Group | Stenfilcon A First, Then Etafilcon A | Etafilcon A First, Then Stenfilcon A
Started | 22; 44 EYES | 19; 38 EYES
Completed | 22; 44 EYES | 19; 38 EYES
Not Completed | 0; 0 EYES | 0; 0 EYES
Period: Lens 2
Arm/Group | Stenfilcon A First, Then Etafilcon A | Etafilcon A First, Then Stenfilcon A
Started | 22; 44 EYES | 19; 38 EYES
Completed | 22; 44 EYES | 19; 38 EYES
Not Completed | 0; 0 EYES | 0; 0 EYES

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Total participants enrolled
Arm/Group | Overall Study
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Comfort
Description: Wearing comfort (throughout the day) for stenfilcon A and etafilcon A toric lens pair is assessed. Scale 0-10, 0= extremely uncomfortable cannot wear at all, 10=very comfortable and feel no lens at all
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Groups:
- Stenfilcon A: Participants randomized to wear stenfilcon A toric lens pair (either first or second) for two weeks during the cross over study.
  stenfilcon A: contact lens
- Etafilcon A Toric: Participants randomized to wear etafilcon A lens pair (either first of second) for two weeks during the cross over study.
  etafilcon A: contact lens
Arm/Group | Stenfilcon A | Etafilcon A Toric
Number analyzed (Participants) | 41 | 41
Number analyzed (eyes) | 82 | 82
units on a scale | 8.2 (2.0) | 7.4 (2.4)

2. Primary Outcome: Dryness
Description: Dryness (throughout the day) for stenfilcon A and etafilcon A toric lens pair is assessed. Scale 0-10, 0=extremely dried and cannot wear lens, 10=feel no dryness at all
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Groups:
- Etafilcon A: Participants randomized to wear etafilcon A toric lens pair (either first or second) for two weeks during the cross over study.
  etafilcon A: contact lens
Arm/Group | Stenfilcon A | Etafilcon A
Number analyzed (Participants) | 41 | 41
Number analyzed (eyes) | 82 | 82
units on a scale | 8.0 (2.0) | 7.4 (2.2)

3. Primary Outcome: Clarity of Vision
Description: Clarity of vision (throughout the day) for stenfilcon A and etafilcon A toric lens pair is assessed. Scale 0-10, 0=blur vision and cannot see at all, 10=very clear with no blur vision at all
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Stenfilcon A | Etafilcon A
Number analyzed (Participants) | 41 | 41
Number analyzed (eyes) | 82 | 82
units on a scale | 8.5 (1.9) | 7.8 (2.4)

4. Primary Outcome: Stability of Vision
Description: Stability of vision (throughout the day) for stenfilcon A and etafilcon A toric lens pair is assessed. Scale 0-10, 0=unstable vision and cannot see at all, 10=always stable vision
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Groups:
- Etafilcon A: Participants randomized to wear etafilcon A toric lens pair (either first of second) for two weeks during the cross over study.
  etafilcon A: contact lens
Arm/Group | Stenfilcon A | Etafilcon A
Number analyzed (Participants) | 41 | 41
Number analyzed (eyes) | 82 | 82
units on a scale | 8.6 (1.8) | 8.0 (2.2)

5. Primary Outcome: Lens Handling
Description: Lens handling for stenfilcon A and etafilcon A toric lens pair is assessed. Scale 0-10, 0=cannot handle at all, 10=no problem at all
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Stenfilcon A | Etafilcon A
Number analyzed (Participants) | 41 | 41
Number analyzed (eyes) | 82 | 82
units on a scale
  At Insertion | 8.8 (1.8) | 7.6 (2.5)
  At Removal | 7.2 (2.9) | 8.9 (1.9)

6. Primary Outcome: Overall Satisfaction
Description: Overall satisfaction for stenfilcon A and etafilcon A toric lens pair is assessed. scale 0-10, 0=extremely un-satisfy, 10=very satisfy
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Stenfilcon A | Etafilcon A
Number analyzed (Participants) | 41 | 41
Number analyzed (eyes) | 82 | 82
units on a scale | 8.1 (2.0) | 7.2 (2.5)

ADVERSE EVENTS:
Time Frame: 2 weeks for each round of lens wear.
Description: Adverse events were assessed for during the follow-up study visits.
Groups:
- Stenfilcon A: Participants randomized to wear stenfilcon A lens pair either as first or second pair in this crossover study.
- Etafilcon A: Participants randomized to wear etafilcon A lens pair either as first or second pair in this crossover study.
Arm/Group | Stenfilcon A | Etafilcon A
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/41
Other Adverse Events (participants affected / at risk) | 0/41 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure restriction on the PI is that the sponsor should be notified of any results communications and has ability to review.